CLINICAL TRIAL: NCT04540133
Title: Dexamethasone Solution and Dexamethasone in Mucolox™ for the Treatment of Oral Inflammatory Ulcerative Diseases
Brief Title: Dexamethasone Solution and Dexamethasone in Mucolox™
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-32068
Record Dates: First submitted 2020-08-28; First posted 2020-09-07 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Oral Lichen Planus; Mucous Membrane Pemphigoid; Pemphigus Vulgaris; Chronic Graft-versus-host-disease
MeSH Terms: conditions — Lichen Planus, Oral; Pemphigoid, Benign Mucous Membrane; Pemphigus; Bronchiolitis Obliterans Syndrome | interventions — Dexamethasone; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dexamethasone 0.5mg/5ml solution in Mucolox™ (group A) (Experimental): Dexamethasone solution (0.5mg/5ml) in Mucolox™ three times a day (TID) swish and spit for 4 weeks
  Interventions: Drug: dexamethasone 0.5mg/5ml solution in Mucolox™
- dexamethasone 0.5mg/5ml solution (Arm B) (Active Comparator): Dexamethasone solution (0.5mg/5ml) TID swish and spit for 4 weeks
  Interventions: Drug: dexamethasone 0.5mg/5ml solution

INTERVENTIONS:
Drug: dexamethasone 0.5mg/5ml solution — Patient with oral ulcerative conditions will be asked to rinse with dexamethasone 0.5mg/5ml solution three times a day for 4 weeks and expectorate
  Other Names: dexamethasone
  Arms: dexamethasone 0.5mg/5ml solution (Arm B)
Drug: dexamethasone 0.5mg/5ml solution in Mucolox™ — Patient with oral ulcerative conditions will be asked to rinse with dexamethasone 0.5mg/5ml solution in Mucolox™ three times a day for 4 weeks and expectorate
  Other Names: dexamethasone solution in Mucolox™
  Arms: dexamethasone 0.5mg/5ml solution in Mucolox™ (group A)

SUMMARY:
Topical steroid therapy is considered the first line of treatment for Oral Inflammatory Ulcerative Diseases with current treatment regimens requiring multiple application or rinses daily. Using Mucolox™ as a vehicle to deliver topical dexamethasone to the oral mucosa has the potential to effectively prolong contact time between the medication. The primary objective of this study is to determine the clinical efficacy and tolerability of compound dexamethasone at 0.5 mg/5 mL in Mucolox™ for the treatment of Oral Inflammatory Ulcerative Diseases as measured by a reduction in oral symptoms between patients treated with compounded dexamethasone 0.5mg/5ml solution in Mucolox™ (group A) and patients treated with topical commercial dexamethasone 0.5mg/5ml solution only (group B). and mucosa, leading to improved clinical outcomes due to the need for less frequent application.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* Patients with symptomatic biopsy proven Oral Inflammatory Ulcerative Diseases (worst VAS sensitivity score ≥ 7 over the last week).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients already on topical or systemic steroids.
* Inability to comply with study instructions.
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
* VAS sensitivity score < 7.
* Pregnant women. A urine pregnancy test will be performed for women of child bearing potential.
* Allergy to fluconazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-12-26 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Villa, DDS, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Sol Silverman Oral Medicine Clinic - UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Final results will be submitted for publication on a peer reviewed journal

REFERENCES:
- [Derived] Lodolo M, Thanasuwat B, Veluppillai P, Bassani G, Villa A. Dexamethasone solution and dexamethasone in Mucolox for the treatment of oral inflammatory ulcerative diseases: A phase II randomized clinical trial. J Oral Pathol Med. 2023 Oct;52(9):860-866. doi: 10.1111/jop.13471. Epub 2023 Aug 7. PMID 37549933

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone 0.5mg/5ml Solution in Mucolox™ (Group A): Dexamethasone solution (0.5mg/5ml) in Mucolox™ three times a day (TID) swish and spit for 4 weeks
  dexamethasone 0.5mg/5ml solution in Mucolox™: Patient with oral ulcerative conditions were asked to rinse with dexamethasone 0.5mg/5ml solution in Mucolox™ three times a day for 4 weeks and expectorate
- Dexamethasone 0.5mg/5ml Solution (Arm B): Dexamethasone solution (0.5mg/5ml) TID swish and spit for 4 weeks
  dexamethasone 0.5mg/5ml solution: Patient with oral ulcerative conditions were asked to rinse with dexamethasone 0.5mg/5ml solution three times a day for 4 weeks and expectorate
Period: Overall Study
Arm/Group | Dexamethasone 0.5mg/5ml Solution in Mucolox™ (Group A) | Dexamethasone 0.5mg/5ml Solution (Arm B)
Started | 15 | 14
Completed | 14 | 14
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone 0.5mg/5ml Solution in Mucolox™ (Group A) | Dexamethasone 0.5mg/5ml Solution (Arm B) | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Median (Full Range); unit: years] | 58 [30 to 79] | 67 [18 to 78] | 58 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 5 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Oral Pain Scores on the Visual Analog Scale (VAS) at 4 Weeks
Description: Oral Pain Scores were measured on the Visual Analog Scale (VAS), the score ranges from 0-10, zero indicating no pain and 10 indicating the worst pain. The pain score measured on a VAS scale will be compared between group A and group B to detect any significant differences pre and post treatment at 4 weeks.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexamethasone 0.5mg/5ml Solution in Mucolox™ (Group A) | Dexamethasone 0.5mg/5ml Solution (Arm B)
Number analyzed (Participants) | 14 | 14
score on a scale | 6.3 (2.4) | 4.4 (3.3)

2. Secondary Outcome: Mean Change From Baseline in Reticulation/Keratosis, Erythema, and Ulceration (REU) Scores at 4 Weeks
Description: Oral lesions were scored using the REU (reticulation,erythema and ulcer) system (form 0 till 49.5). Reticulations were scored from 0 to 1 (0 = no white striations, 1 = presence of white striations or keratotic papules); erythematous lesions from 0 to 3 by area of involvement (0 = no lesion, 1 = lesions less than 1 cm2, 2 = lesions from 1 to 3 cm2, 3 = lesions greater than 3 cm2); ulcers from 0 to 3 by area of involvement. The higher is the score the more severe is the disease. In order to evaluate the clinical improvement in clinician-reported outcome measures for oral lesions, REU scores within the compound dexamethasone solution in Mucolox™ group (Arm A) will be compared to that in the dexamethasone solution only group (Arm B). The REU scores will be summarized descriptively for each arm at pre-treatment, post-treatment, and pre-to-post treatment change. The pre-to-post treatment change will be compared between the arms using either student's t-test o
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexamethasone 0.5mg/5ml Solution in Mucolox™ (Group A) | Dexamethasone 0.5mg/5ml Solution (Arm B)
Number analyzed (Participants) | 14 | 14
score on a scale | 2.5 (3.1) | 3.2 (1.7)

ADVERSE EVENTS:
Time Frame: 1 month (study period)
Arm/Group | Dexamethasone 0.5mg/5ml Solution in Mucolox™ (Group A) | Dexamethasone 0.5mg/5ml Solution (Arm B)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT04540133/Prot_SAP_001.pdf